CLINICAL TRIAL: NCT01620047
Title: Postoperative Knee Strength Following Total Knee Replacement: A Double-Blinded Randomized Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Tampa General Hospital (Other)
Responsible Party: Principal Investigator, Enrico Camporesi, President, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TGH-007 IRB # Pro00002055
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-09

CONDITIONS: Total Knee Replacement; Primary Knee Arthroplasty
Keywords: Regional Anesthesia; Post-operative pain management; Femoral Nerve Block; Total Knee Replacement
MeSH Terms: interventions — Fentanyl; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Femoral Nerve Fentanyl (Experimental): Fentanyl 3 µg/ml delivered continuously through a femoral nerve sheath catheter for 24 hours post-total knee replacement. All study drugs were continuously infused for a 24 hour period at a basal rate of 10ml/hour starting from the time the patient entered the post anesthesia care unit (PACU).
  Interventions: Drug: Fentanyl
- Femoral Nerve Ropivacaine (Active Comparator): Ropivacaine 0.1% continuously delivered through a femoral nerve sheath catheter for 24 hours post-total knee replacement. All study drugs were continuously infused for a 24 hour period at a basal rate of 10ml/hour starting from the time the patient entered the post anesthesia care unit (PACU).
  Interventions: Drug: Ropivacaine
- Intravenous Fentanyl with placebo (Placebo Comparator): Control group which received 0.9% normal saline delivered through a femoral nerve sheath catheter in addition to a continuous intravenous infusion of fentanyl 3 µg/ml via a PCA pump. All study drugs were continuously infused for a 24 hour period at a basal rate of 10ml/hour starting from the time the patient entered the post anesthesia care unit (PACU).
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl 3 µg/ml continuously infused for a 24 hour period at a basal rate of 10ml/hour starting from the time the patient entered the post anesthesia care unit (PACU)through a femoral nerve sheath catheter.
  Arms: Femoral Nerve Fentanyl
Drug: Ropivacaine — Ropivacaine 0.1% delivered through a femoral nerve sheath catheter continuously for a 24 hour period at a basal rate of 10ml/hour starting from the time the patient entered the post anesthesia care unit (PACU).
  Arms: Femoral Nerve Ropivacaine
Drug: Fentanyl — 0.9% normal saline delivered through a femoral nerve sheath catheter in addition to a continuous intravenous infusion of fentanyl 3 µg/ml via a PCA pump for a 24 hour period at a basal rate of 10ml/hour starting from the time the patient entered the post anesthesia care unit (PACU).
  Arms: Intravenous Fentanyl with placebo

SUMMARY:
Major surgery involving the knee is often associated with severe postoperative pain. Postoperative pain control remains a significant contributor to delayed recovery and length of hospital stay. Approaches to minimize postoperative pain after surgery are a matter of major concern due to the need for early mobilization, a crucial factor in good postoperative rehabilitation. Femoral nerve blocks by either continuous infusion or single injection of anesthetics provide an effective method for analgesia while minimizing the need for systemic opioid therapy, reducing the opioid induced side effects, and facilitating early ambulation. Administration of fentanyl has shown to be a highly effective method to control pain after Total Knee Replacement (TKR). The investigators hypothesize that fentanyl infusions will result in greater post-operative strength in the operative knee.

DETAILED DESCRIPTION:
All subjects scheduled to receive a unilateral, primary total knee replacement were evaluated for eligibility in the preoperative anesthesia center. Adults, older than 18 years of age, ASA I-III were included in the study. Subjects who were either pregnant, on anticoagulant therapy, allergic to opioids, local anesthetics, chronic pain patients, history of traumatic lower extremity injury, or had a body mass index of greater than 35 kg/m2 were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary total knee replacement
* ASA class I-III
* 18 years and older

Exclusion Criteria:

* Patient refusal
* Pregnancy
* Coagulopathy
* Adverse/allergic reaction to any opioids or local anesthetics
* History of long-term opioid use (greater than 60 days)
* Infection
* Traumatic lower extremity injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devanand Mangar, MD, Principal Investigator — Florida Gulf-to-Bay Anesthesiology Associates LLC
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

REFERENCES:
- [Background] Charous MT, Madison SJ, Suresh PJ, Sandhu NS, Loland VJ, Mariano ER, Donohue MC, Dutton PH, Ferguson EJ, Ilfeld BM. Continuous femoral nerve blocks: varying local anesthetic delivery method (bolus versus basal) to minimize quadriceps motor block while maintaining sensory block. Anesthesiology. 2011 Oct;115(4):774-81. doi: 10.1097/ALN.0b013e3182124dc6. PMID 21394001
- [Background] Bauer M, Wang L, Onibonoje OK, Parrett C, Sessler DI, Mounir-Soliman L, Zaky S, Krebs V, Buller LT, Donohue MC, Stevens-Lapsley JE, Ilfeld BM. Continuous femoral nerve blocks: decreasing local anesthetic concentration to minimize quadriceps femoris weakness. Anesthesiology. 2012 Mar;116(3):665-72. doi: 10.1097/ALN.0b013e3182475c35. PMID 22293719
- See also: American Society of Anesthesiology — http://asahq.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, randomized, double-blinded study performed between April and November 2011. Patients were recruited in the pre-operative clinic 3 to 7 days prior to undergoing a total knee replacement.
Groups:
- Intravenous Fentanyl: Control group which received 0.9% normal saline delivered through a femoral nerve sheath catheter in addition to a continuous intravenous infusion of fentanyl 3 µg/ml via a PCA pump. All study drugs were continuously infused for a 24 hour period at a basal rate of 10ml/hour starting from the time the patient entered the post anesthesia care unit (PACU).
Period: Overall Study
Arm/Group | Femoral Nerve Fentanyl | Femoral Nerve Ropivacaine | Intravenous Fentanyl
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Nerve Fentanyl | Femoral Nerve Ropivacaine | Intravenous Fentanyl With Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 8 | 8 | 21
  >=65 years | 15 | 12 | 12 | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 69 (9) | 67 (12) | 67 (9) | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 14 | 38
  Male | 9 | 7 | 6 | 22
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Postoperative Strength (Extension)
Description: To assess extension force postoperatively to discern differences in muscle strength retention between continuous femoral nerve sheath catheter administration of fentanyl or Ropivacaine or a continuous IV infusion of fentanyl.
Time Frame: 24 hours post-surgery
Population: Per protocol
Measure: Median (Full Range); unit: Nm/kg
Arm/Group | Femoral Nerve Fentanyl | Femoral Nerve Ropivacaine | Intravenous Fentanyl With Placebo
Number analyzed (Participants) | 20 | 20 | 20
Nm/kg | .08 [0.01 to 0.28] | .03 [0.01 to 0.17] | .05 [0 to 0.13]

2. Secondary Outcome: VAS Scores and Postoperative Supplemental Morphine Consumption
Description: Secondary Objective
  * To determine the amount of required supplemental analgesia during the postoperative period.
  * To determine postoperative analgesia using a Visual Analog Scale (VAS) 0 - 10 centimeter line.
Time Frame: 24 hours post-surgery
Reporting Status: Not Posted

3. Secondary Outcome: Serum Fentanyl Levels
Description: To identify a difference in serum fentanyl levels among the groups.
Time Frame: 24 hours post-surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Femoral Nerve Fentanyl | Femoral Nerve Ropivacaine | Intravenous Fentanyl With Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 5/20 | 10/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Femoral Nerve Fentanyl (N=20) | Femoral Nerve Ropivacaine (N=20) | Intravenous Fentanyl With Placebo (N=20)
Nausea (Gastrointestinal disorders) | 9 | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No